CLINICAL TRIAL: NCT07009652
Title: Proposal for the Organisation of the Procedure for Extracorporeal Cardiopulmonary Resuscitation of Patients With Sudden Cardiac Arrest in the Pre-hospital Environment of the Moravian-Silesian Region
Brief Title: Optimization of Transport and Use of a Mobile ECMO Team in Patients With Sudden Cardiac Arrest in the Moravian-Silesian Region
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Emergency Medical Services, Moravian-Silesian Region (Unknown)
Responsible Party: Sponsor
Other Study IDs: CEPR-01-ECPR
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest With Successful Resuscitation; Cardiac Arrest, Cause Unspecified
Keywords: cardiac arrest; extracorporeal membrane oxygenation; out-of-hospital cardiac arrest; extracorporeal cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECPR and ECMO: Patients undergoing extracorporeal cardiopulmonary resuscitation (ECPR).
  Interventions: Procedure: Extracorporeal cardiopulmonary resuscitation (ECPR)

INTERVENTIONS:
Procedure: Extracorporeal cardiopulmonary resuscitation (ECPR) — Extracorporeal cardiopulmonary resuscitation (commonly known as ECPR) is a method of cardiopulmonary resuscitation (CPR) that passes the patient's blood through a machine in a process to oxygenate the blood supply.

SUMMARY:
This study evaluates the feasibility of implementing a mobile extracorporeal membrane oxygenation (ECMO) team and optimizing patient transport logistics.

DETAILED DESCRIPTION:
The aim of the study is to improve neurological outcomes in out-of-hospital cardiac arrest (OHCA) cases in the Moravian-Silesian Region. By analysing regional epidemiological and demographic data, the project aims to identify key factors for reducing the time from collapse to the initiation of ECMO and to support the development of effective protocols for extracorporeal cardiopulmonary resuscitation (ECPR).

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest
* indication for ECPR

Exclusion Criteria:

* death at the scene of the accident
* withdrawal of the informed consent

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients indicated for ECPR after out-of-hospital cardiac arrest, for whom transport of the patient to an ECMO centre or deployment of an ECMO team is logistically manage-able.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome after 30 days (CPC score) | 30 days
  Assessment of the neurological status of patients 30 days after the event using the Cerebral Performance Category (CPC) scale, which measures the extent of neurological impairment:
  * CPC 1 = good neurological condition
  * CPC 2 = mild impairment
  * CPC 3-5 = serious impairment, vegetative state or death The primary endpoint of the study is the proportion of patients with a favourable neurological outcome (CPC 1-2).

SECONDARY OUTCOMES:
Time from collapse to initiation of ECMO | Up to 2 hours
  Measuring the time (in minutes) from patient collapse to ECMO initiation. The aim is to analyse how this time affects neurological outcome.
Transport time to the ECMO centre | Up to 2 hours
  Measurement of the time (in minutes) from the arrival of the Emergency Medical Services (EMS) at the scene to the admission of the patient to the ECMO centre.
Arrival time for the mobile ECMO team to the scene | Up to 2 hours
  Time interval (in minutes) from activation of the mobile ECMO team to its arrival at the scene. The aim is to evaluate the effectiveness of the model and the potential time benefit of intervention in the field.

CONTACTS AND LOCATIONS:
Overall Officials: Nela Walachová, Mgr., Principal Investigator — University Hospital Ostravs
Locations (2):
- Czechia (2):
  - Emergency Medial Services, Moravian-Silesian Region, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.